CLINICAL TRIAL: NCT01800305
Title: A Randomized, Positive-controlled, Single-dose, Dose-escalation Phase I Trial to Evaluate Safety & Tolerability, and Explore the Pharmacokinetics and Pharmacodynamics Profile of Pegylated rhEPO in Male Healthy Individual
Brief Title: PK & PD Study of Pegylated rhEPO, and Evaluated Its Safety and Tolerability in Male Healthy Individual
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TB1209EPO
Record Dates: First submitted 2013-02-24; First posted 2013-02-27 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: PK & PD study; rhEPO; Pegylated rhEPO; male healthy subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegylated rhEPO (Experimental): Subcutaneous single-dose administration of 0.5mcg/kg, 1.0mcg/kg, 1.6 mcg/kg, 2.4 mcg/kg, 3.2 mcg/kg，3.2mcg/kg, 4.2mcg/kg, 5.5 mcg/kg, 7.2 mcg/kg, 9.3 mcg/kg (in dose-escalation, if the previous dose is confirmed to be safe.started with the second 3.2mcg/kg dose,Every subject takes Niferex 150mg every day, from day 1 to day 20. ) of the test drug (Pegylated rhEPO)
  Interventions: Drug: Pegylated rhEPO
- EPIAO® (Active Comparator): Subcutaneous six-dose administration of 50IU/kg or 150IU/kg, as randomization, of the comparator drug(EPIAO®) at day 1, 3, 5, 8, 10, 12.
  Interventions: Drug: EPIAO®

INTERVENTIONS:
Drug: Pegylated rhEPO
  Arms: Pegylated rhEPO
Drug: EPIAO®
  Arms: EPIAO®

SUMMARY:
The object of this randomized, parallel, positive controlled study is to explore the pharmacokinetics and pharmacodynamics profile of the test drug after single-dose subcutaneous administration, compared to the comparator drug (EPIAO®) after multiple-dose subcutaneous administration, by assessing plasma concentration of the drug and the reticulocyte count, hemoglobin concentration and hematocrit following subcutaneous administration, evaluate the security and tolerability of the test drug in healthy subjects, and provide sufficient information for dose selection in the future phase II and III study.

ELIGIBILITY:
Inclusion Criteria:

* Agree to all the purposes of the study by signing and dating the informed consent.
* Male, aged between 18 and 40 years, age disparity of each group should less than 10 years.
* Body weight ≥ 50kg, and body mass index (BMI) between 18 kg/m2 and 26kg/m2 at screening.
* Hemoglobin between 131g/L and 162g/L, hematocrit between 41% and 49%, and reticulocyte between 0.5% and 2%.
* Transferrin saturation and serum ferritin are in the normal range.
* Physical condition: vital signs, physical examination and laboratory tests ( including routine blood, biochemical tests, coagulation indicators, serum folic acid, vitamin B12, urine test, HBsAg, anti-HCV, anti-HIV, Immunoglobulin (IgA, IgM, IgG), thyroid function (T3, T4, TSH), autoantibodies), chest-X-ray, 12-lead ECG should all in normal range, or without significant clinically abnormal.

Exclusion Criteria:

* Presence of organic disease in heart, liver, kidney, brain; or presence of cardiovascular, pulmonary, gastrointestinal, urinary, neurological, endocrine, immunity, genitourinary or other systems disease.
* Subjects with familial genetic disease, mental illness, or physical disability.
* History of drug allergy.
* Orthostatic hypotension, systolic blood pressure <90mmHg.
* Habitual medication, including Chinese herbal medicine.
* Poor inclusion conditions (e.g. infirm).
* Smoker (smoke everyday or more than 7 cigarettes per week)，alcoholics (more than 40g/day, equivalent to 100ml/day of 50 degree of white spirit).
* Participate in any other drug trials as the subjects within the previous 3 months.
* As blood donated within the previous 3 months, or experienced massive blood loss due to trauma or surgery.
* Other conditions which in the opinion of the investigator precluding enrollment into the study (e.g. poor compliance).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Serum concentration of rhEPO | 0 hour before drug administration and 1, 3, 6, 9, 12, 14, 16, 24, 36, ,48, 72, 96, 120, 144, 168, 192, 216,240, 264, 288, 300, 312, 360, 408, 480, 648, 984,1320 hour after drug administration
  * Time frame of day 12 for comparator drug: 0 hour before drug administration and 1, 3, 6, 9, 14, 16 hour after last dose administration.
  * For comparator drug, blood collection of 0, 48, 96, 168, 216, and 264 hour should before drug administration.
Plasma reticulocyte count | 0 hour before and 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 360, 408, 480, 648,984,1320 hour after first drug administration.
  For comparator drug, blood collection of 48, 96, 168, 216, and 264 hour should before drug administration
Plasma hemoglobin concentration | 0 hour before and 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 360, 408, 480, 648,984,1320 hour after first drug administration.
  For comparator drug, blood collection of 48, 96, 168,216, and 264 hour should before drug administration
Plasma hematocrit | 0 hour before and 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 360, 408, 480, 648,984,1320 hour after first drug administration.
  For comparator drug, blood collection of 48, 96, 168,216, and 264 hour should before drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhenman, Ph.D, Principal Investigator — Beijing 302 Hospital
Locations (1):
- 302 Military Hospital of China, Beijing, China